CLINICAL TRIAL: NCT00224913
Title: NMES for Older Individuals After Total Knee Arthroplasty
Brief Title: Electrical Stimulation After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Center for Medical Rehabilitation Research (NCMRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01HD041055 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-10-12 (Estimated); Status verified 2005-10

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: osteoarthritis; quadriceps; inhibition; functional outcome; electrical stimulation
MeSH Terms: conditions — Osteoarthritis; Inhibition, Psychological

INTERVENTIONS:
Procedure: Neuromuscular electrical stimulation
Procedure: Voluntary exercise

SUMMARY:
Total knee arthroplasty (TKA) is performed more than 300,000 times a year in the United States, most often for osteoarthritis (OA). While pain is predictably reduced, function does not typically ever reach that of age-matched, uninjured subjects. Quadriceps weakness has been implicated in the development and progression of knee OA and is a significant problem after TKA. Voluntary exercise has been ineffective at restoring quadriceps strength after TKA. The aims of this study are: 1) to assess the effectiveness of high-level neuromuscular electrical stimulation as an adjunct to ongoing intensive, early rehabilitation in restoring quadriceps strength and improving the functional outcome after primary TKA, and 2) to identify the physiological and morphological bases for improvements in quadriceps strength and functional outcome.

DETAILED DESCRIPTION:
Reduced muscle strength from illness or injuries often leads to loss of function and independence in the elderly. The recovery of muscle strength and function in disabled elderly individuals is a major challenge in rehabilitation. The etiology of the muscle weakness with injury or age is not fully elucidated. Training programs designed to maximize strength gains in young individuals may not be optimal in the elderly because the cause of the weakness and the morphology of the muscle may be different for young vs. old people. The overall goal of this work is to determine if physiologically and morphologically based rehabilitation programs are more effective than traditional rehabilitation to counter changes in muscle strength and function in older individuals. Neuromuscular electrical stimulation (NMES) may be used to improve strength and function following injury or surgery. This study provides motivation for exploring the use of NMES with the elderly. We posit that using NMES to augment a traditional rehabilitation program for elderly patients with osteoarthritis following total knee arthroplasties (TKA) will result in greater strength and functional gains than using only traditional rehabilitation. Elderly patients with osteoarthritis who undergo TKAs serve as ideal subjects for testing the effectiveness of rehabilitation programs become those patients almost always exhibit marked quadriceps weakness that is resistant to traditional physical rehabilitation. More than 300,000 TKAs are performed each year in the United States to treat osteoarthritis of the knee in older individuals. So, the successful rehabilitation of elder patients following TKA is an important and challenging problem. The specific aims of this proposal are: 1) To assess the effectiveness of high-level neuromuscular electrical stimulation is an adjunct to ongoing intensive, early rehabilitation in restoring quadriceps strength and improving the functional outcome after primary TKA, and 2) To identify the physiological and morphological bases for improvements in quadriceps strength and functional outcome

A total of 200 subjects will participate in this study. Functional and strength testing provides information for the patients' clinical treatment and allow us to monitor their progress. This information will also help in the design of a training program for individuals following a total knee replacement that optimizes the return to full level of function after surgery. MRI screening will provide information regarding the size of the thigh muscle at various periods throughout rehabilitation. It will enable us to assess the impact of post-operative treatment on increasing the size of the thigh muscle. Patients will be asked to participate in functional and strength testing sessions, lasting about 1½ hours, at the following times: 0-2 weeks before surgery, 3-4 weeks, 6-7 weeks, 10-12 weeks, 6 months, 1 year, and 2 years after surgery. MRI testing will last about 30 minutes per session and will be performed 0-2 weeks before surgery, and 3-4 weeks, 10-12 weeks, and 1 year after surgery.

Functional testing will include 5 parts: a timed walking test, a timed stair climbing test, a timed balance test, a timed step test, and a six-minute walk test. A strength test will be used to assess the strength of the thigh muscles.

The second part of this study involves treatment. Patients participate in 6 weeks of physical therapy, 3 times per week. They are randomly assigned to one of 2 groups. One group will participate in a traditional rehabilitation program. The other group will receive electrical stimulation for strengthening of the thigh muscle in addition to the traditional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* TKA for unilateral tricompartmental knee OA

Exclusion Criteria:

* Insulin dependent diabetes
* neurological conditions
* other lower extremity orthopedic problems that affect function
* BMI>40

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-03

PRIMARY OUTCOMES:
Quadriceps Strength
Quadriceps Activation
Functional Tests

SECONDARY OUTCOMES:
Self reports of function

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Snyder-Mackler, PT, ScD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

REFERENCES:
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Result] Mizner RL, Snyder-Mackler L. Altered loading during walking and sit-to-stand is affected by quadriceps weakness after total knee arthroplasty. J Orthop Res. 2005 Sep;23(5):1083-90. doi: 10.1016/j.orthres.2005.01.021. Epub 2005 Mar 28. PMID 16140191
- [Result] Mizner RL, Petterson SC, Snyder-Mackler L. Quadriceps strength and the time course of functional recovery after total knee arthroplasty. J Orthop Sports Phys Ther. 2005 Jul;35(7):424-36. doi: 10.2519/jospt.2005.35.7.424. PMID 16108583
- [Result] Stevens JE, Mizner RL, Snyder-Mackler L. Neuromuscular electrical stimulation for quadriceps muscle strengthening after bilateral total knee arthroplasty: a case series. J Orthop Sports Phys Ther. 2004 Jan;34(1):21-9. doi: 10.2519/jospt.2004.34.1.21. PMID 14964588
- [Result] Stevens JE, Mizner RL, Snyder-Mackler L. Quadriceps strength and volitional activation before and after total knee arthroplasty for osteoarthritis. J Orthop Res. 2003 Sep;21(5):775-9. doi: 10.1016/S0736-0266(03)00052-4. PMID 12919862
- [Result] Mizner RL, Stevens JE, Snyder-Mackler L. Voluntary activation and decreased force production of the quadriceps femoris muscle after total knee arthroplasty. Phys Ther. 2003 Apr;83(4):359-65. PMID 12665406
- [Derived] Laufer Y, Snyder-Mackler L. Response of male and female subjects after total knee arthroplasty to repeated neuromuscular electrical stimulation of the quadriceps femoris muscle. Am J Phys Med Rehabil. 2010 Jun;89(6):464-72. doi: 10.1097/PHM.0b013e3181dd8c0e. PMID 20489392
- [Derived] Petterson SC, Mizner RL, Stevens JE, Raisis L, Bodenstab A, Newcomb W, Snyder-Mackler L. Improved function from progressive strengthening interventions after total knee arthroplasty: a randomized clinical trial with an imbedded prospective cohort. Arthritis Rheum. 2009 Feb 15;61(2):174-83. doi: 10.1002/art.24167. PMID 19177542